CLINICAL TRIAL: NCT05121792
Title: Web Based Therapist and Patient Tutorials on Prolonged Grief. Study 1
Brief Title: Web Based Therapist Tutorial on Prolonged Grief
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Center for Psychological Consultation (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Katherine Shear, MD, Marion E. Kenworthy Professor of Psychiatry, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AAAT7389 Study1; 1R41MH118126-01A1 (NIH)
Record Dates: First submitted 2021-11-05; First posted 2021-11-16 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Prolonged Grief Disorder
Keywords: grief; therapy; training
MeSH Terms: conditions — Prolonged Grief Disorder

STUDY DESIGN:
Intervention Model Description: Study 1 is an open-label (non-randomized) study to generate pilot data on effectiveness, and to evaluate feasibility and acceptability of the therapist online training program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Therapist online training in Prolonged Grief Disorder Therapy (Experimental): Participants will be given access to an online 10-module interactive tutorial about Prolonged Grief Disorder Therapy.
  Interventions: Behavioral: Web Based Therapist Tutorial on Prolonged Grief Disorder Therapy

INTERVENTIONS:
Behavioral: Web Based Therapist Tutorial on Prolonged Grief Disorder Therapy — The tutorial consists of 10 online modules following the main procedures of the Prolonged Grief Disorder Therapy (formerly known as Complicated Grief Treatment). Each module includes didactic information and interactive activities and videos, and takes approximately 30 minutes to review. Participants can study the material at their own pace.

SUMMARY:
Death of a loved one is a difficult life experience. About 1 in 10 bereaved people are strongly affected by the loss and grieve intensely for a long time. As a result of the COVID-19 pandemic, more people may struggle with grief. The investigators have developed and tested a talk therapy for prolonged grief.

The investigators have developed an online grief training for clinicians. The investigators will test if clinicians benefit from the online training and if they find it helpful and engaging. The investigators will recruit 30 mental health professionals as trainees to undergo the training. The mental health professionals will complete questionnaires before and after training to determine how much they learned and how much they liked the training.

DETAILED DESCRIPTION:
The investigators developed a short-term, manualized Prolonged Grief Disorder Therapy (PGDT), originally known as Complicated Grief Treatment and found it efficacious in three large National Institute of Mental Health (NIMH) sponsored randomized controlled trials. Facilitating access to training in Empirically Based Treatments has been identified as a national priority by both mental health professional organizations and NIMH. One way to help disseminate therapist training on EBT of Prolonged Grief Disorder (PGD) is through the use of new technologies. The investigators recently developed an online therapist training program in PGDT and a patient facing therapist-assisted web-based form of PGDT. The investigators are now looking to evaluate the acceptability and effectiveness of each of these online tools in pilot studies.

The tutorial contains 10 modules, each about 20-40 minutes long with information needed for effective delivery of PGDT. Participants will be encouraged to space out the tutorial vs. taking it in a few long sessions, to facilitate knowledge retention. A post-test will be given immediately after completing each module, as testing done closer to when the material was learned also improves retention. Participants will be encouraged to complete the tutorial within 5 weeks (about one hour or two modules per week). Consistent with continuing education guidelines, successful completion will require an overall score of 80% on post-tests. Participants would need to retake the module until a passing score is obtained. Interactive Patient Scenarios will be integrated into the tutorial at strategic points, in order to integrate conceptual and applied knowledge. All participants will be asked to evaluate whether the stated learning goals of each module were met and complete user satisfaction questionnaires on both the technical aspects of the on-line tutorial (using the System Usability Scale), and the clinical content (using the User Satisfaction Questionnaire). Participants will have access to the tutorial indefinitely, in order to provide a resource that they can refer back to as they begin to use these skills with patients.

ELIGIBILITY:
Inclusion Criteria:

* Mental health professional

Exclusion Criteria:

* Student or employee of Columbia University

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2021-10-28 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
User Satisfaction Questionnaire (USQ) | Week 5 (after training completion)
  The USQ evaluates participant satisfaction with the clinical content of web-based applications, and how effective the participant felt the learning was. The USQ contains 15 statements, each rated on a 4-point scale (strongly agree, agree, disagree, strongly disagree), and covers several dimensions of the user experience. It also solicits open-ended feedback. The scale ranges from 15 to 60, with a higher score indicating user satisfaction. The investigators will consider an overall mean score of 45 (i.e., an average score of 3 ["agree" on all items]) to demonstrate acceptable user satisfaction with the clinical content.
System Usability Scale (SUS) | Week 5 (after training completion)
  The SUS is a 10-item self-report scale designed to evaluate the usability and user satisfaction with web-based and other technologies. It obtains quantitative feedback on a 0-100 scale regarding the effectiveness, efficiency, and satisfaction users experience while interacting with engineered systems. A mean SUS score significantly greater than 50.9 (mean rating for systems considered "Okay") would be evidence of system user-friendliness; "Good" is considered a mean rating of 71.4 or better.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth A. Kobak, PhD, Principal Investigator — Center for Psychological Consultation, WI; Katherine Shear, MD, Principal Investigator — Columbia School of Social Work
Locations (2):
- United States (2):
  - Center for Complicated Grief, Columbia School of Social Work, New York, New York
  - Center for Psychological Consultation, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shear K, Frank E, Houck PR, Reynolds CF 3rd. Treatment of complicated grief: a randomized controlled trial. JAMA. 2005 Jun 1;293(21):2601-8. doi: 10.1001/jama.293.21.2601. PMID 15928281
- [Background] Shear MK, Reynolds CF 3rd, Simon NM, Zisook S, Wang Y, Mauro C, Duan N, Lebowitz B, Skritskaya N. Optimizing Treatment of Complicated Grief: A Randomized Clinical Trial. JAMA Psychiatry. 2016 Jul 1;73(7):685-94. doi: 10.1001/jamapsychiatry.2016.0892. PMID 27276373
- [Derived] Kobak K, Shear MK, Skritskaya NA, Bloom C, Bottex G. A Web-Based Therapist Training Tutorial on Prolonged Grief Disorder Therapy: Pre-Post Assessment Study. JMIR Med Educ. 2023 Mar 27;9:e44246. doi: 10.2196/44246. PMID 36972105